CLINICAL TRIAL: NCT02498899
Title: Message 2: The Effect of Message Content and Clinical Outcome on Patient's Perception of Physician Compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-0279; NCI-2015-01553 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Video; Questionnaires; Surveys
MeSH Terms: interventions — Surveys and Questionnaires; Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video 1 + Questionnaires (Experimental): Participants complete 4 questionnaires at baseline. Participants then watch a short video. At end of video, 3 questionnaires completed. Participants then read a small story about the patient in the video. Afterwards, another set of questionnaires completed.
  Interventions: Behavioral: Questionnaires; Behavioral: Video
- Video 2 + Questionnaires (Experimental): Participants complete 4 questionnaires at baseline. Participants then watch a short video. At end of video, 3 questionnaires completed. Participants then read a small story about the patient in the video. Afterwards, another set of questionnaires completed.
  Interventions: Behavioral: Questionnaires; Behavioral: Video

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete questionnaires at baseline, after watching a video, and after reading a story about the patient in the video.
  Other Names: Surveys
Behavioral: Video — Participants watch a video lasting about 4 minutes.

SUMMARY:
The goal of this research study is to learn how patients view their doctor's compassion about supportive care and treatment options for advanced cancer patients.

DETAILED DESCRIPTION:
If you agree to take part in this study, during an already scheduled office visit, you will complete the following:

* Basic information about you will be collected from your medical record (such as your date of birth, date of diagnosis, sex, and religion).
* You will complete 4 questionnaires about any symptoms you may be having, how hopeful you are in general, how you are dealing with the disease, your trust in the medical profession, and your strength of religious faith. It should take about 10 minutes total to complete all questionnaires.

You will then be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Each group will watch a short video that shows actors playing a doctor and patient having a conversation about different cancer treatment options. Each video is about 4 minutes long and will discuss the same material, but the message shown in the videos will be different for each group.

After you watch the video, you will complete 3 questionnaires that will ask about your impression of the doctor in the video, how hopeful you think the doctor was, if you think the doctor was professional, and how you would rate the doctor overall. It should take about 8 minutes total to complete all questionnaires.

You will then read a small story about the patient in the video. Afterwards, you will complete the same 3 questionnaires that you filled out after you watched the video. You will also complete an additional questionnaire about your impression of the doctor's compassion and trustworthiness. This should take less than 10 minutes to complete.

Length of Study:

It should take about 25 minutes total to watch the video and to complete all questionnaires. Your active participation on this study will be over after you have completed the last questionnaire.

Other Information:

You are taking part in this study alone. Your family members will not be in the room with you. If you request, your family may be able remain in the room, but the investigators ask that they remain silent.

This is an investigational study.

Up to 128 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced cancer, defined as locally advanced, recurrent or metastatic disease
2. Follow up patients seen in the outpatient Supportive Care Center.
3. Age >/= 18 years-old
4. English speaking

Exclusion Criteria:

1. Altered cognitive status as determined by the interviewer based on the ability to understand the nature of the study and consent process.
2. Patients suffering from a severe psychiatric disorder or condition that would significantly interfere with study participation, as determined by the Principal Investigator or by the attending palliative care physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Rating of Physician's Compassion | 1 day
  Participant's rating of physician's compassion scored by using a 5-item tool consisting of five 0-10 numerical rating scales assessing five dimensions: warm-cold, pleasant-unpleasant, compassionate-distant, sensitive insensitive, caring-uncaring. Sum of the five scales gives a final score representing physician's compassion with a 0 to 50 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberson C. Tanco, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org